CLINICAL TRIAL: NCT02533011
Title: Heparin Binding Protein (HBP) in Sepsis for the Prediction of Disease Progression
Brief Title: Evaluation of the Heparin Binding Protein Levels in Sepsis
Acronym: HBP
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 602986
Record Dates: First submitted 2015-07-16; First posted 2015-08-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Sepsis; Infection; Septic Shock
Keywords: Sepsis; Heparin Binding Protein
MeSH Terms: conditions — Sepsis; Infections; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 24 Hours: HBP lab test performed 24 hours after meeting sepsis inclusion criteria.
  Interventions: Other: HBP lab test
- 48 Hours: HBP lab test performed 48 hours after meeting sepsis inclusion criteria.
  Interventions: Other: HBP lab test
- 72 Hours: HBP lab test performed 72 hours after meeting sepsis inclusion criteria.
  Interventions: Other: HBP lab test

INTERVENTIONS:
Other: HBP lab test — Plasma level of Heparin Binding Protein will be evaluated on extra blood specimens already collected as part of standard of care.
  Other Names: Plasma level of heparin binding protein

SUMMARY:
Present criteria used to define sepsis are non-specific, making it difficult to both distinguish sepsis from other diseases and to predict which patients are likely to become more severely ill. In standard care, patients at risk of becoming more severely ill are neither identified nor indicated for resuscitative efforts until they develop hemodynamic insufficiency or organ failure; after progression to severe disease, mortality increases significantly. The identification of risk patients can lead to earlier initiation of resuscitation therapies and potentially lead to reduced morbidity and mortality. This study aims to determine whether Heparin-binding protein (HBP), which is secreted from neutrophils during infection and a mediator of vascular leakage, can act as a biomarker for the progression to severe sepsis with circulatory failure.

The objective of this study is to validate the utility of HBP to predict the development of delayed onset organ dysfunction in sepsis in patients and to compare the performance of HBP relative to currently used prognostic biomarkers in sepsis.

DETAILED DESCRIPTION:
Sepsis is a heterogeneous disorder caused by an invasive infection that results in host inflammatory response. The underlying pathogenesis is complex and dependent on the etiologic microorganism, site of infection, and host factors. Present criteria defining sepsis (including change of body temperature, increased heart and respiration rates, and leukocytosis/leukopenia) are non-specific making it difficult to distinguish sepsis from other diseases and in particular to predict which patients are likely to become more severely ill. The consensus definition of sepsis has been debated over the past years and one suggested approach is to focus more on the presence of organ dysfunction. In standard care, patients at risk of becoming more seriously ill are not identified nor indicated for resuscitative efforts until they develop hemodynamic insufficiency or organ failure. However, after progression to severe disease mortality increases significantly. A recent study showed that almost a quarter of patients presenting with uncomplicated sepsis in an Emergency Department (ED) developed severe sepsis or septic shock within 72 hours. Delayed in-hospital progression to increased organ dysfunction was associated with increased transfer to the intensive care unit (ICU) and increased hospital length of stay. The identification of risk patients can lead to earlier initiation of resuscitation therapies and potentially lead to reduced morbidity and mortality. There are also increasing evidence that a single episode of severe sepsis has negative impact on quality of life and mortality several years after the actual incident. Also, recent studies indicate that less severe organ dysfunction, such as small increases in serum creatinine, are associated with increased long-term mortality among sepsis survivors.

Mechanisms that trigger the release of heparin-binding protein (HBP) from neutrophils in the presence of bacteria have previously been reported. HBP has several functions such as a chemo-attractant and as an activator of monocytes and macrophages. Also, it induces vascular leakage by interacting with the capillary endothelium and breaking cell barriers. In vivo studies have demonstrated that HBP released by the complex formed by the group A streptococcal M1 protein and fibrinogen induces a massive tissue edema contributing to severe organ damage. In clinical investigations, the release of HBP has been demonstrated in various infectious diseases caused by a wide array of bacteria. A recent single-center study of patients admitted for suspected infection and fever showed that plasma levels of HBP were significantly higher among patients who presented with or developed severe sepsis with circulatory failure.

A prospective observational study in a tertiary care Emergency Department. Patients must be identified and enrolled within 72 hours of qualifying inclusion criteria. At this time, unused blood samples collected for routine testing will be examined and the plasma level of HBP will be recorded; only blood samples processed by the lab within 3 hours of collection will be used. In addition, physiologic variables detailed in the data elements section, including mental status, metabolic, renal, heme, hepatic, respiratory, cardiovascular, resuscitation, and vasopressor use will be recorded. Patients who meet the inclusion criteria will be identified. Researchers will collect and record a resuscitation summary for a span of 4 hours; this data, outlined in the data elements section, will be linked to the quality improvement (QI) database of Sepsis Research. Additionally, the patient's HBP plasma levels will be measured from unused blood samples collected for routine lab testing time (T) 24, 48, and 72-hours (T24, T48, T72) after meeting the inclusion criteria (T0); resuscitation summaries will also be collected at T24, T48, T72. For patients meeting sepsis alert criteria, T0 will be defined as the time that the patient qualified; those enrolled based on Predisposition, Injury, Response, Organ dysfunction (PIRO) score will have T0 defined as the time hospital admission was ordered. Patients will be followed throughout their time in the hospital and their outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a bacterial or viral infection
* 18 years or older
* Meet the sepsis alert criterion (Hypotension (BP < 90 after 2 L of fluids or lactate ≥ 4) OR
* PIRO (Predispose, Infection, Response, Organ dysfunction ) score ≥ 15 .

Exclusion Criteria:

* Minors (less than 18 years of age)
* Patients who do not meet sepsis criteria as described above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted through the emergency department with infection.
Sampling Method: Non-Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Infection with organ dysfunction, defined as PIRO (Predisposition, Insult, Response, Organ Dysfunction) Score greater than 5 | 72 hours after meeting sepsis criteria
  Patients with septic shock or severe sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C. Arnold, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

REFERENCES:
- [Background] Dremsizov T, Clermont G, Kellum JA, Kalassian KG, Fine MJ, Angus DC. Severe sepsis in community-acquired pneumonia: when does it happen, and do systemic inflammatory response syndrome criteria help predict course? Chest. 2006 Apr;129(4):968-78. doi: 10.1378/chest.129.4.968. PMID 16608946
- [Background] Shapiro N, Howell MD, Bates DW, Angus DC, Ngo L, Talmor D. The association of sepsis syndrome and organ dysfunction with mortality in emergency department patients with suspected infection. Ann Emerg Med. 2006 Nov;48(5):583-90, 590.e1. doi: 10.1016/j.annemergmed.2006.07.007. PMID 17052559
- [Background] Vincent JL, Opal SM, Marshall JC, Tracey KJ. Sepsis definitions: time for change. Lancet. 2013 Mar 2;381(9868):774-5. doi: 10.1016/S0140-6736(12)61815-7. No abstract available. PMID 23472921
- [Background] Glickman SW, Cairns CB, Otero RM, Woods CW, Tsalik EL, Langley RJ, van Velkinburgh JC, Park LP, Glickman LT, Fowler VG Jr, Kingsmore SF, Rivers EP. Disease progression in hemodynamically stable patients presenting to the emergency department with sepsis. Acad Emerg Med. 2010 Apr;17(4):383-90. doi: 10.1111/j.1553-2712.2010.00664.x. PMID 20370777
- [Background] Arnold RC, Sherwin R, Shapiro NI, O'Connor JL, Glaspey L, Singh S, Medado P, Trzeciak S, Jones AE; Emergency Medicine Shock Research Network (EM Shock Net) Investigators. Multicenter observational study of the development of progressive organ dysfunction and therapeutic interventions in normotensive sepsis patients in the emergency department. Acad Emerg Med. 2013 May;20(5):433-40. doi: 10.1111/acem.12137. PMID 23672356
- [Background] Bastani A, Galens S, Rocchini A, Walch R, Shaqiri B, Palomba K, Milewski AM, Falzarano A, Loch D, Anderson W. ED identification of patients with severe sepsis/septic shock decreases mortality in a community hospital. Am J Emerg Med. 2012 Oct;30(8):1561-6. doi: 10.1016/j.ajem.2011.09.029. Epub 2011 Dec 26. PMID 22204997
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Rivers EP, Katranji M, Jaehne KA, Brown S, Abou Dagher G, Cannon C, Coba V. Early interventions in severe sepsis and septic shock: a review of the evidence one decade later. Minerva Anestesiol. 2012 Jun;78(6):712-24. Epub 2012 Mar 23. PMID 22447123
- [Background] Yende S, D'Angelo G, Kellum JA, Weissfeld L, Fine J, Welch RD, Kong L, Carter M, Angus DC; GenIMS Investigators. Inflammatory markers at hospital discharge predict subsequent mortality after pneumonia and sepsis. Am J Respir Crit Care Med. 2008 Jun 1;177(11):1242-7. doi: 10.1164/rccm.200712-1777OC. Epub 2008 Mar 27. PMID 18369199
- [Background] Cuthbertson BH, Elders A, Hall S, Taylor J, MacLennan G, Mackirdy F, Mackenzie SJ; Scottish Critical Care Trials Group; Scottish Intensive Care Society Audit Group. Mortality and quality of life in the five years after severe sepsis. Crit Care. 2013 Apr 16;17(2):R70. doi: 10.1186/cc12616. PMID 23587132
- [Background] Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA; Genetic and Inflammatory Markers of Sepsis (GenIMS) Investigators. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010 Mar;77(6):527-35. doi: 10.1038/ki.2009.502. Epub 2009 Dec 23. PMID 20032961
- [Background] Linder A, Fjell C, Levin A, Walley KR, Russell JA, Boyd JH. Small acute increases in serum creatinine are associated with decreased long-term survival in the critically ill. Am J Respir Crit Care Med. 2014 May 1;189(9):1075-81. doi: 10.1164/rccm.201311-2097OC. PMID 24601781
- [Background] Herwald H, Cramer H, Morgelin M, Russell W, Sollenberg U, Norrby-Teglund A, Flodgaard H, Lindbom L, Bjorck L. M protein, a classical bacterial virulence determinant, forms complexes with fibrinogen that induce vascular leakage. Cell. 2004 Feb 6;116(3):367-79. doi: 10.1016/s0092-8674(04)00057-1. PMID 15016372
- [Background] McNamara C, Zinkernagel AS, Macheboeuf P, Cunningham MW, Nizet V, Ghosh P. Coiled-coil irregularities and instabilities in group A Streptococcus M1 are required for virulence. Science. 2008 Mar 7;319(5868):1405-8. doi: 10.1126/science.1154470. PMID 18323455
- [Background] Macheboeuf P, Buffalo C, Fu CY, Zinkernagel AS, Cole JN, Johnson JE, Nizet V, Ghosh P. Streptococcal M1 protein constructs a pathological host fibrinogen network. Nature. 2011 Apr 7;472(7341):64-8. doi: 10.1038/nature09967. PMID 21475196
- [Background] Linder A, Akesson P, Brink M, Studahl M, Bjorck L, Christensson B. Heparin-binding protein: a diagnostic marker of acute bacterial meningitis. Crit Care Med. 2011 Apr;39(4):812-7. doi: 10.1097/CCM.0b013e318206c396. PMID 21200320
- [Background] Kjolvmark C, Akesson P, Linder A. Elevated urine levels of heparin-binding protein in children with urinary tract infection. Pediatr Nephrol. 2012 Aug;27(8):1301-8. doi: 10.1007/s00467-012-2132-x. Epub 2012 Mar 13. PMID 22410798
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Shapiro NI, Trzeciak S, Hollander JE, Birkhahn R, Otero R, Osborn TM, Moretti E, Nguyen HB, Gunnerson KJ, Milzman D, Gaieski DF, Goyal M, Cairns CB, Ngo L, Rivers EP. A prospective, multicenter derivation of a biomarker panel to assess risk of organ dysfunction, shock, and death in emergency department patients with suspected sepsis. Crit Care Med. 2009 Jan;37(1):96-104. doi: 10.1097/CCM.0b013e318192fd9d. PMID 19050610
- [Background] Reinhart K, Bauer M, Riedemann NC, Hartog CS. New approaches to sepsis: molecular diagnostics and biomarkers. Clin Microbiol Rev. 2012 Oct;25(4):609-34. doi: 10.1128/CMR.00016-12. PMID 23034322